CLINICAL TRIAL: NCT04705662
Title: Investigating the Effects of Iron on the Gastrointestinal Tract in Health.
Brief Title: GI Effects of Iron in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Consultant Clinical Scientist, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FGC-20-002
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Iron Deficiency Anemia Treatment; Microbial Colonization; Iron-deficiency; Iron Deficiency Anemia
Keywords: ferrous sulphate
MeSH Terms: conditions — Communicable Diseases; Anemia, Iron-Deficiency | interventions — Surveys and Questionnaires; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferrous Sulphate (Other): This is a single arm study, all participants will take Ferrous sulphate 200mg (65mg elemental iron) for 4 weeks (+/- 2 days). Participants will be required to take 2 tablets per day.
  Interventions: Diagnostic Test: Lactulose breath test; Other: Stool sample; Other: Daily Diary; Other: Irritable Bowel syndrome severity scoring system (IBS-SSS) questionnaire; Dietary Supplement: Ferrous Sulphate

INTERVENTIONS:
Diagnostic Test: Lactulose breath test — Participants will complete a 3 hour breath test pre and post iron supplementation. This will include taking 4 exploratory samples for volatile organic compound (VOC) analysis.
Other: Stool sample — Participants will provide a stool sample pre and post iron supplementation
Other: Daily Diary — Monitoring stool form, consistency and frequency on a daily basis
Other: Irritable Bowel syndrome severity scoring system (IBS-SSS) questionnaire — Participants will complete the questionnaire pre and post iron supplementation
Dietary Supplement: Ferrous Sulphate — Participants will take Ferrous sulphate 200mg (65mg elemental iron) for 4 weeks (+/- 2 days). Participants will be required to take 2 tablets per day.

SUMMARY:
Over recent years there has been a lot of research looking at how the bacteria in our gut affects our health. Some medications are known to cause changes in gut bacteria.

Many patients that are prescribed iron report gastrointestinal side effects. This research project aims to see if the cause of the gastrointestinal side effects is due to iron causing changes in the gut bacteria. This can be detected via measuring the levels of hydrogen and methane and other compounds in the breath and stool.

DETAILED DESCRIPTION:
Iron deficiency anaemia is the most common health issue worldwide, with approximately >1.2 billion people affected. In the UK, iron deficiency anaemia most commonly affects pre-school aged children and women aged 15-49 years. In 2011, an estimated 14% of non-pregnant, and 23% of pregnant women in the UK had iron deficiency anaemia, and 2-5% of male and post-menopausal women were also affected. Whilst compared to other areas of the world IDA has a mild public health significance to the UK, it can be the reason for up-to 13% of referrals to gastroenterologists.

Treating IDA with oral supplements or IV infusions are both effective at restoring bodily iron stores. However, success is often greater in those receiving their iron intravenously, due to frequent non-adherence to oral tablets as a result of their side effects. Gastrointestinal complaints, most commonly constipation, are reported by up to 60% of people that take oral iron supplements. These GI complaints causes up to 50% of patient to not follow their treatment plan, meaning their iron deficiency anaemia persists. However, patients that receive intravenous iron infusions instead do not report these symptoms. This suggests that oral iron has an impact on the GI tract as intravenous iron will bypass the gastrointestinal lumen but the mechanism of this remains uncertain.

To investigate the side effects of oral iron supplements and research a potential mechanism for the cause of iron supplement side effects, this study will require healthy volunteers to take ferrous sulphate for 4 weeks. Pre and post intervention participants will be required to provide a stool sample, complete a breath test and answer questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Participant is a male or non-pregnant female (confirmed by pregnancy test) and is age 18 years to 60 years.
3. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.
4. Participant has capacity to understand written English.
5. Participant has no significant medical diagnosis or current or previous chronic gastrointestinal disease requiring medication or surgery (apart from appendectomy). Participant has no disease that would contraindicate iron supplementation e.g. haemochromatosis.
6. Participant is not on regular prescription medicines unless a stable dose for the past 6-months and duration of the trial.
7. Participant has a body mass index (BMI) of 18.5 - 34.9 kg/m2 (bounds included).
8. Participant agrees to follow pre-test diet for 24 hours before giving test sample.
9. Participant agrees to refrain from strenuous physical activity on the day of the breath test.
10. Participant agrees to refrain from smoking on the day of the breath test.
11. Participant agrees to an overnight fast on the night before the breath test. Food and drink must be withheld until after all breath test samples have been taken.
12. Participant agrees to not take any probiotic for 14 days before the breath test or during the study.
13. Participant has not taken antibiotics for 4-weeks before the start of the study or during the study

Exclusion Criteria:

1. Participant has no significant medical diagnosis or current or previous chronic gastrointestinal disease requiring medication or surgery (apart from appendectomy). Participant has no disease that would contraindicate iron supplementation e.g. haemochromatosis.
2. Participant is pregnant or breast feeding.
3. Participant takes medication known to impact the gut microbiome:

   1. Antibiotics used in the last 4 weeks
   2. Regular use of laxatives or anti-diarrheal medication
4. Participant is taking a regular prescription medication that has a contraindication with oral iron supplementation.
5. Participant has undergone a colonoscopy/sigmoidoscopy in the 1 week prior to enrolment.
6. Participant regularly consumes probiotics, prebiotics, fibre supplements in the 4 weeks prior to enrolment and/or is unwilling to exclude the use of probiotics from the diet during the study period.
7. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or sponsor member.
8. Participant has had previous abdominal or colorectal surgery except appendectomy or hysterectomy.
9. Participant has had oral iron supplementation of IV iron supplementation in the 12 months prior to enrolment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Breath methane levels | 4 weeks apart
  Difference in methane levels in breath samples from baseline and 4-weeks since commencing iron therapy. This will be measured in parts per million (ppm).

SECONDARY OUTCOMES:
Volatile organic compounds (VOC) in breath | 4 weeks apart
  Difference in any breath gas markers. This is exploratory so will look to see what is present at baseline and see how it changes over the 4 week study period.
Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | 4 weeks apart
  Comparison in change of IBS-SSS score from baseline to 4 weeks since commencing iron therapy. The minimum score is 0 and maximum score is 500. The greater the score, the worse the severity and frequency of symptoms of abdominal pain and distention, and increased dissatisfaction of overall bowel functioning.
Stool consistency via the Bristol Stool Chart | 4 weeks apart
  Change in stool frequency and form according to the bristol stool chart scale from baseline to 4 weeks since commencing iron therapy.
Gut Microbiome analysis via stool samples | 4 weeks
  Qualitative and Quantitative data for faecal microorganisms at baseline and 4-weeks since commencing iron therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, Study Chair — The Functional Gut Clinic
Locations (2):
- United Kingdom (2):
  - The Functional Gut Clinic, Cambridge, Greater Manchester
  - The Functional Gut Clinic, Manchester, Greater Manchester

IPD SHARING:
Plan to Share IPD: No
Results will be written up and published in journal articles and presented at conferences